CLINICAL TRIAL: NCT06766656
Title: Comparison of Transverse and Longitudinal Incisions for Venous Access Port Placement
Acronym: port placement
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Tomasz Skladzien, Senior Lecturer, Jagiellonian University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1072.6120.115.2024
Record Dates: First submitted 2025-01-04; First posted 2025-01-09 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-01

CONDITIONS: Central Venous Access Devices; Implantable Venous Access Port
Keywords: Implantable venous access port (IVAP), Comfort, Complications; Central venous access devices

STUDY DESIGN:
Intervention Model Description: Vessel cannulation is performed percutaneously using an ultrasound machine and fluoroscopy. The "pocket" for the vascular port is made through a small incision in the skin in the subclavicular area. The skin incision can be made transversely or longitudinally, depending on the preferences of the physician performing the procedure. In both cases, this does not affect the further course of the procedure. Both methods of creating a vascular "pocket" are commonly used. The procedures are performed as part of one-day stays, and after the procedure, patients are discharged home.
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- transversely incision (Active Comparator): The "pocket" for the vascular port is made through a small incision in the skin in the subclavicular area. The skin incision will be made transversely
  Interventions: Procedure: Incision
- longitudinally incision (Active Comparator): The "pocket" for the vascular port is made through a small incision in the skin in the subclavicular area. The skin incision will be made longitudinally,
  Interventions: Procedure: Incision

INTERVENTIONS:
Procedure: Incision — The "pocket" for the vascular port is made through a small incision in the skin in the subclavicular area. The skin incision can be made transversely or longitudinally

SUMMARY:
The aim of the study is to assess whether the direction of skin incision affects pain within the first 24 hours, patient comfort 7 days after the procedure, procedure time, and the occurrence of early complications related to vascular port implantation.

DETAILED DESCRIPTION:
The vascular port implantation procedure is used in patients who require long-term access to veins, e.g. during chemotherapy, long-term drug administration or blood collection. This procedure is performed under local anesthesia, by cannulating the internal jugular vein - left or right and making an incision to place the port on the chest wall (so-called "pocket") in the subclavicular area on the side of the cannulated vein.

Vessel cannulation is performed percutaneously using an ultrasound machine and fluoroscopy. The "pocket" for the vascular port is made through a small incision in the skin in the subclavicular area. The skin incision can be made transversely or longitudinally, depending on the preferences of the physician performing the procedure. In both cases, this does not affect the further course of the procedure. Both methods of creating a vascular "pocket" are commonly used. The procedures are performed as part of one-day stays, and after the procedure, patients are discharged home.

To the best of our knowledge, this is the first study that will compare the direction of the skin incision. In our study, we wanted to compare pain in the first 24 hours, patient comfort after 7 days of the procedure, procedure time, occurrence of early complications related to vascular port implantation. Patients undergoing the vascular port implantation procedure will be divided into two groups, one will have a transverse incision, and the other a longitudinal incision in order to place the port in the subcutaneous tissue. Patients will receive a questionnaire to fill out (in the appendix to the application) and will have their pain monitored on the NRS scale at 1, 2, 6, 12, 24 hours after the procedure. Additionally, on the 7th day after the procedure, I will be asked to assess any discomfort associated with the presence of the vascular port on a scale of 0-5. Data will be collected by phone. Additionally, we will measure the procedure time and occurrence of any complications related to port implantation.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria:

Age > 18 and < 80 years Informed consent Need for central venous access port implementation under local anesthesia

Exclusion Criteria:

Impaired blood clotting Ongoing antiplatelet drugs therapy, except acetylsalicylic acid Trauma or surgical past history on both shoulder girdles Known central venous thrombosis (subclavian vein, upper vena cava) Known pneumothorax Chronic opioid use Septic state Agranulocytosis

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Pain | 1 day
  pain monitored on the NRS scale at 1, 2, 6, 12, 24 hours after the procedure

SECONDARY OUTCOMES:
Discomfort | 7 days
  discomfort associated with the presence of the vascular port on a scale of 0-5

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Intensive Interdisciplinary Care, Collegium Medicum, Jagiellonian University, Krakow, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Erdemir A, Rasa HK. Impact of central venous port implantation method and access choice on outcomes. World J Clin Cases. 2023 Jan 6;11(1):116-126. doi: 10.12998/wjcc.v11.i1.116. PMID 36687176
- [Result] Walser EM. Venous access ports: indications, implantation technique, follow-up, and complications. Cardiovasc Intervent Radiol. 2012 Aug;35(4):751-64. doi: 10.1007/s00270-011-0271-2. Epub 2011 Sep 16. PMID 21922348